CLINICAL TRIAL: NCT05092308
Title: Perspectives of Parents About Their Infants' Sleep: What do the Mothers Wish? What do the Fathers Think?
Brief Title: Perspectives of Parents About Their Infants' Sleep
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 09.2021.719
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Insomnia
Keywords: sleep; insomnia; children; actigraphy; marital relationship
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents and their children with Behavioral insomnia: Parents and their children aged 6-36 months with sleep problems will be invited to participate into the study from Sleep Outpatient Clinic
- Parents and their children without sleep problem: Parents and their children aged 6-36 months without sleep problems will be invited to participate into the study followed up in Well Child Clinic

SUMMARY:
Behavioral insomnia of childhood (BIC) is a common problem in early infancy. The whole family is affected by the problem, but research usually relies only on maternal perception and report. This mixed-method study aimed to explore maternal and paternal perspectives about their child's sleep and sleep problems in early childhood. Secondly, infants' sleep will be measured objectively with actigraphy. Parental mental health, marital relationship and sleep will be evaluated in order to explore the effects on the perception of their infant's sleep.

DETAILED DESCRIPTION:
Sleep is essential for healthy growth and development of children. Behavioral insomnia of childhood is reported as a common sleep problem of early childhood with a prevalence of 26-68% according to the definition and study population.

Behavioral insomnia of childhood not only affects children's health but also has impacts on parental mental health and family functioning. Most studies on early childhood sleep problems rely on maternal report. However, both parents are affected by children's sleep problem. It is therefore essential for pediatric healthcare professional to understand both mothers' and fathers' perception and interpretation of their children's sleep and sleep problems in the context of family and culture to suggest culturally appropriate intervention according to the family's needs.

This study is designed to thematically analyze maternal and paternal perspectives of their child's sleep and sleep problems in early childhood.

Parents of children aged 6-36 months with and without sleep problems will be invited to participate into the study. Both parents of 10-15 children applying for sleep problems to Sleep Outpatient Clinic and both parents of 10-15 children followed up in Well Child Clinic without sleep problems will be included from October 2021 to June 2022. Semi-structured individual in depth interviews will be conducted with both mothers and fathers but in different sessions separately to explore parental views and perception of their child's sleep and sleep problems. The interviews are expected to last between 30-45 minutes and will be audio-recorded and transcribed for thematic analysis. Through these interviews the investigators will learn what kind of differences are present between the parents' perspectives of infants with and without sleep problems.

Sleep of all children will be evaluated by Turkish version of the expanded brief infant sleep questionnaire, actigraphy and sleep diary. Sociodemographic information will be collected. Parents in patient and control group will be assessed for the confounding factors by Patient Health Questionnaire-9, Generalized Anxiety Scale-7 test, Relationship Satisfaction Scale, Marital Life Satisfaction Scale and Pittsburgh Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria:

* Parents and their 6-36 months old children

Exclusion Criteria:

* Divorced or separated couples
* Infants less than 37 weeks of gestational age
* Children with diagnosed developmental problems

Ages: 6 Months to 36 Months | Sex: All
Age Groups: Child
Study Population: - Parents and their 6-36 months old children with and without sleep problems
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Perspectives of parents on infant sleep | Baseline
  The semi- structured individual interviews will be conducted with mothers and fathers of infants with and without sleep problems. Both parents of an infant will be interviewed in different sessions to detect any discrepancies between their opinions. The topic guide will include parental views, perceptions and interpretations of their infants' sleep and expectations regarding interventions.

SECONDARY OUTCOMES:
Parental anxiety | Baseline
  • Parental anxiety will be measured with Generalized anxiety scale-7. It is a seven item scale developed to screen for anxiety in general in primary care settings. The questionnaire score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. Cut off score for Turkish validation has been set at 8.
• Parental depression symptoms | Baseline
  • Parental depression symptoms will be measured with Patient Health Questionnaire-9. It is a nine item scale used to screen for the presence and severity of depressive symptoms. As a severity measure, the PHQ-9 score ranges from 0 to 27, with each of the nine items scored from 0 (not at all) to 3 (nearly every day). A score of 10 or above indicates depressive disorder. Turkish validation has been done.
• Global relationship | baseline
  • Global relationship will be measured with Relationship Assessment Scale. This is a brief measure of global relationship satisfaction, which consists of seven items, each rated on a five-point Likert scale, ranging from 1 (not well), to 5 (very well). The scale is suitable to use with any individuals who are in an intimate relationship such as married couples or cohabiting couples.
• Married-life satisfaction scale | baseline
  • Married-life satisfaction scale is a 5-item scale developed to measure married life satisfaction. Higher scores indicate better marital satisfaction.
Parental Sleep quality | Baseline
  • Parental sleep quality will be measured with Pittsburgh sleep quality index. It is a questionnaire which assesses sleep disturbances over a 1-month time interval. If the PUKI global score is greater than 5, it indicates poor sleep quality. Turkish validation has been done.
Infant sleep wake patterns | Baseline
  • Infants sleep wake patterns will be measured with actigraphy. Actigraphy is a wrist-watch like device that continuously measures motion and estimates sleep-wake patterns by measuring motion in natural settings. It is a valid method to objectively assess infants' sleep. Sleep wake patterns will be assessed by Philips Respironics Mini-Mitter Actiwatch-2 for 3 days at home environment and sleep diaries within 5-minute intervals will be filled out by parents simultaneously. The following actigraphic sleep metrics will be used: 1) wake after sleep onset (WASO); 1) sleep of latency (SOL); and 3) number of awakenings (NW), sleep duration, sleep efficiency.
Infant sleep parameters | Baseline
  • Infant sleep parameters will be measured by Expanded-Brief Infant Sleep Questionnaire (BISQ) :BISQ is a screening questionnaire for sleep in infants and young children. Variables include nocturnal sleep duration, daytime sleep duration, number of night awakenings, duration of night time wakefulness, nocturnal sleep onset time, settling time, method of falling asleep, location of sleep. If the child woke up more than 3 times per night, spent more than 1 hour in wakefulness during the night, or spent less than 9 hours in sleep (day and night), then they were considered as poor sleepers

IPD SHARING:
Plan to Share IPD: Undecided
Requests for wider sharing of data (for example in response to information on Marmara University webpages and in publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate and meets the criteria set by the university; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.